CLINICAL TRIAL: NCT05931237
Title: Evaluation of the Inter-individual Variability Associated With the Interaction Between Flavan-3-ols From Cranberry and Gut Microbiota - an Exploratory Study
Brief Title: Cranberry Flavan-3-ols Consumption and Gut Microbiota in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Symrise (Industry)
Responsible Party: Principal Investigator, Yves Desjardins, Full professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Metacann
Record Dates: First submitted 2023-06-07; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cranberry extract capsules (PREBIOCRAN(TM)) (Experimental): Cranberry extract capsules consumed twice a day providing 82.3 mg of flavan-3-ols daily.
  Interventions: Dietary Supplement: Cranberry extract capsules

INTERVENTIONS:
Dietary Supplement: Cranberry extract capsules — Cranberry extract capsules (Prebiocran(TM))
  Other Names: Prebiocran cranberry extract

SUMMARY:
Consumption of (poly)phenols is recognized to have beneficial effects on health. However, heterogeneous results are obtained in clinical trials due to high inter-individual variability. The objective of this pilot study is to characterize the inter-individual variability associated with the interaction of (poly)phenols from cranberry and gut microbiota.

The participants (n=39) of this study are healthy adults aged between 23 and 63 years old and consumed cranberry extract rich in (poly)phenols for 4 days. Plasma, urine and feces were collected to quantify gut microbial (poly)phenols metabolites and to profile the fecal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Stable weight
* Stable or no medication
* Stable diet
* Stable physical activity

Exclusion Criteria:

* Pregnant women
* Antibiotic and/or probiotic use three months prior to the study
* Smokers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Targeted metabolomic assessment (UPLC-QToF-MS) of the change in gut microbial flavan-3-ols metabolites concentration in 24h urine before and after supplementation of a cranberry extract. | Change from Baseline concentration in flavan-3-ols gut metabolites at 4 days
  Determine the change in concentration of flavan-3-ols metabolites generated by the gut microbial metabolism before and after the consumption of 82.3 mg/day of cranberry extract in 24h urine samples (µmol/24h). The following microbial metabolites of flavan-3-ols will be determined by UPLC-QToF-MS: 5-(3´-hydroxyphenyl)-γ-valerolactone (3-HPVL), 5-(3´,4´-dihydroxyphenyl)-γ-valerolactone (3,4-DHPVL), 5-(3´-hydroxyphenyl)valeric acid (3-HPVA),and 5-(3´,4´-dihydroxyphenyl)valeric acid (3,4-DHPVA), 1-(3',4'-Dihydroxyphenyl)-3-(2",4",6"-trihydroxyphenyl)-propan-2-ol (3,4-DHPP-2-ol), 1-(3'-Hydroxyphenyl)-3-(2",4",6"-trihydroxyphenyl)-propan-2-ol (3-HPP-2-ol), 3-(3',4'-Dihydroxyphenyl)propanoic acid (3,4-DHPPA), and 3-(3'-Hydroxyphenyl)propanoic acid (3-HPPA).
Targeted metabolomic assessment (UPLC-QToF-MS) of the change in gut microbial flavan-3-ols metabolites concentration in plasma before and after supplementation of a cranberry extract. | Change from Baseline concentration in flavan-3-ols gut metabolites at 4 days
  Determine the change in concentration of flavan-3-ols metabolites generated by the gut microbial metabolism before and after the consumption of 82.3 mg/day of cranberry extract in plasma samples (nmol/L). The following microbial metabolites of flavan-3-ols will be determined by UPLC-QToF-MS: 5-(3´-hydroxyphenyl)-γ-valerolactone (3-HPVL), 5-(3´,4´-dihydroxyphenyl)-γ-valerolactone (3,4-DHPVL), 5-(3´-hydroxyphenyl)valeric acid (3-HPVA),and 5-(3´,4´-dihydroxyphenyl)valeric acid (3,4-DHPVA), 1-(3',4'-Dihydroxyphenyl)-3-(2",4",6"-trihydroxyphenyl)-propan-2-ol (3,4-DHPP-2-ol), 1-(3'-Hydroxyphenyl)-3-(2",4",6"-trihydroxyphenyl)-propan-2-ol (3-HPP-2-ol), 3-(3',4'-Dihydroxyphenyl)propanoic acid (3,4-DHPPA), and 3-(3'-Hydroxyphenyl)propanoic acid (3-HPPA).
Targeted metabolomic assessment (UPLC-QToF-MS) of the change in gut microbial flavan-3-ols metabolites concentration in fecal samples before and after supplementation of a cranberry extract. | Change from Baseline concentration in flavan-3-ols gut metabolites at 4 days
  Determine the change in concentration of flavan-3-ols metabolites generated by the gut microbial metabolism before and after the consumption of 82.3 mg/day of cranberry extract in fecal samples (nmol/g). The following microbial metabolites of flavan-3-ols will be determined by UPLC-QToF-MS: 5-(3´-hydroxyphenyl)-γ-valerolactone (3-HPVL), 5-(3´,4´-dihydroxyphenyl)-γ-valerolactone (3,4-DHPVL), 5-(3´-hydroxyphenyl)valeric acid (3-HPVA),and 5-(3´,4´-dihydroxyphenyl)valeric acid (3,4-DHPVA), 1-(3',4'-Dihydroxyphenyl)-3-(2",4",6"-trihydroxyphenyl)-propan-2-ol (3,4-DHPP-2-ol), 1-(3'-Hydroxyphenyl)-3-(2",4",6"-trihydroxyphenyl)-propan-2-ol (3-HPP-2-ol), 3-(3',4'-Dihydroxyphenyl)propanoic acid (3,4-DHPPA), and 3-(3'-Hydroxyphenyl)propanoic acid (3-HPPA).

SECONDARY OUTCOMES:
Change in the gut microbiota composition before and after supplementation of a cranberry extract. | Change from Baseline microbial composition at 4 days
  Determine the effect of a 4-day supplementation of cranberry extract on the composition of the gut microbiota through 16S ribosomal ribonucleic acid (rRNA) sequencing. Evaluate the changes in composition of the major microbial families and genus of participants' fecal samples. Changes in microbiota functional profile will be assessed by comparing over and under-expressed Amplicon Sequence Variants (ASV) against the SILVA databased based on the Kyoto Encyclopedia of Genes and Genomes (KEGG) Ontology (KO) functional and pathway profiles.
Targeted metabolomic assessment (UPLC-QToF-MS) of the change in short-chain fatty acids (SCFA) concentration in 24h urine before and after supplementation of a cranberry extract. | Change from Baseline SCFA at 4 days
  Determine the effect of a 4-day cranberry extract supplementation on the changes in concentration (nmol/24h) in SCFA (acetate, propionate, butyrate, valerate), in 24h urine samples (UPLC-QToF-MS).
Targeted metabolomic assessment (UPLC-QToF-MS) of the change in bile acids concentration in plasma before and after supplementation of a cranberry extract. | Change from Baseline bile acids at 4 days
  Determine the effect of a 4-day cranberry extract supplementation on the changes in bile acids (cholic acid, chenodeoxycholic acid, ursodeoxycholic acid, lithocholic) concentration in plasma samples (nmol/L) (UPLC-QToF-MS).
Targeted metabolomic assessment (UPLC-QToF-MS) of the change in tryptophan metabolites concentration in fecal samples before and after supplementation of a cranberry extract. | Change from Baseline tryptophan metabolites at 4 days
  Determine the effect of a 4-day cranberry extract supplementation on the changes in tryptophan metabolites (serotonin, kynurenine, tryptamine, quinolinic acid) concentration in fecal samples (nmol/g) (UPLC-QToF-MS).
Targeted metabolomic assessment (UPLC-QToF-MS) of the change in short-chain fatty acids (SCFA) concentration in the plasma before and after supplementation of a cranberry extract. | Change from Baseline SCFA at 4 days
  Determine the effect of a 4-day cranberry extract supplementation on the changes in concentration (nmol/24h) in SCFA (acetate, propionate, butyrate, valerate), in plasma samples (nmol/L)(UPLC-QToF-MS).
Determine the effect of a 4-day cranberry extract supplementation on the changes in bile acid concentration in fecal samples (UPLC-QToF-MS). | Change from Baseline bile acids at 4 days
  Determine the effect of a 4-day cranberry extract supplementation on the changes in bile acids (cholic acid, chenodeoxycholic acid, ursodeoxycholic acid, lithocholic) concentration in fecal samples (nmol/g) (UPLC-QToF-MS).

CONTACTS AND LOCATIONS:
Locations (1):
- Laval University, Québec, Canada

IPD SHARING:
Plan to Share IPD: No